CLINICAL TRIAL: NCT00234975
Title: Evaluation of Clinical Response and Safety in HIV Positive Subjects Co-infected With Hepatitis C Treated With a Kaletra Containing HAART Regimen
Brief Title: Safety of Lopinavir/Ritonavir (Kaletra) in HIV/HCV Co-infected Subjects vs Baseline Liver Biopsy Metavir Score
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PUER-02-003
Record Dates: First submitted 2005-09-13; First posted 2005-10-10 (Estimated); Last update posted 2013-01-03 (Estimated); Status verified 2013-01

CONDITIONS: HIV Infection
Keywords: Lopinavir; Ritonavir; Phase 4; HIV
MeSH Terms: conditions — HIV Infections | interventions — Lopinavir; Ritonavir; lopinavir-ritonavir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HCV + (Active Comparator)
  Interventions: Drug: Lopinavir/Ritonavir
- HCV - (Active Comparator)
  Interventions: Drug: Lopinavir/Ritonavir

INTERVENTIONS:
Drug: Lopinavir/Ritonavir — 400 mg/ 100 mg BID. Both arms use Kaletra 400/100 mg BID, plus NRTI chosen by the investigator
  Other Names: ABT-378, lopinavir/ritonavir, Kaletra

SUMMARY:
The purpose of this study is to evaluate clinical response and safety of a Kaletra containing antiretroviral treatment regimen in HIV positive subjects with HCV coinfection.

ELIGIBILITY:
Inclusion Criteria:

* Documented HIV positive.
* At least 18 years of age.
* Does not exhibit evidence of acute illness (especially any acute liver disease, except hepatitis C)
* Subject has not been treated for an active opportunistic infection within 30 days of the baseline visit.
* Subject Has a Karnofsky Score greater than or equal to 70.
* Subject does not require and agrees not to take, for the duration of the study, any of the following medications that are contraindicated with Kaletra: astemizole, terfenadine, midazolam, triazolam, cisapride, certain ergot derivatives (ergotamine, dihydroergotamine, ergonovine, and methylergonovine), pimozide, propafenone and flecainide. Rifampin, a potent enzyme inducer, should not be administered with the study medication, because of the possibility of significant decreases in Kaletra concentration during concurrent administration.
* The subject agrees not to take any medication, including over-the-counter medicine, alcohol, recreational drugs or herbal preparations without the knowledge and permission of the principal investigator.
* Subject had laboratory testing within the previous three months and the most recent testing demonstrates all of the following: Hemoglobin> 8.0 g/dL; absolute neutrophil count > 750 cells/mL; Platelet count > 20,000/mL; ALT or AST </=10 x upper limit of normal (ULN); Creatinine< 1.5 x ULN; Triglycerides </=750 mg/dL.
* Subjects have no evidence of grade III or IV adverse event or laboratory abnormality (except for LFTs).

Exclusion Criteria:

No exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2002-10; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Primary Outcome Measure | Baseline, Week 4, Week 8, Week 16 and Week 24
  Changes in liver functions enzyme.

SECONDARY OUTCOMES:
Secondary Outcome Measures | Baseline, Week 4, Week 8, Week 16 and Week 24
  Changes in HIV viral load, CD4/CD8 cell count, and Hepatitis C viral load

CONTACTS AND LOCATIONS:
Overall Officials: Carlos R Rivera-Vazquez, MD, Study Director — AbbVie
Locations (11):
- Puerto Rico (11):
  - Site Reference ID/Investigator# 4118, Bayamón
  - Site Reference ID/Investigator# 4119, Bayamón
  - Site Reference ID/Investigator# 6298, Juana Díaz
  - Site Reference ID/Investigator# 6284, Las Piedras
  - Site Reference ID/Investigator# 4101, Mayagüez
  - Site Reference ID/Investigator# 4116, Playa de Ponce
  - Site Reference ID/Investigator# 4117, Ponce
  - Site Reference ID/Investigator# 4099, Ponce
  - Site Reference ID/Investigator# 4086, Rio Piedras
  - Site Reference ID/Investigator# 4080, San Juan
  - Site Reference ID/Investigator# 4100, Santurce

REFERENCES:
- See also: Related Info — http://rxabbvie.com